CLINICAL TRIAL: NCT01341717
Title: Open-labelled, Randomized, Active-controlled, Parallel-arm, Single-center Study on Effect of Sitagliptin on T2DM Patients on Treatment With Metformin and Insulin
Brief Title: Effects of Sitagliptin on Type 2 Diabetes Mellitus Patients on Treatment With Metformin and Insulin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jothydev's Diabetes and Research Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JDC/SITA/021/2011
Record Dates: First submitted 2011-04-23; First posted 2011-04-26 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Sitagliptin; Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Sitagliptin Phosphate; glimepiride; Metformin; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sitagliptin along with metformin and insulin (Experimental)
  Interventions: Drug: Sitagliptin; Drug: Glimepiride; Drug: Metformin; Drug: Insulin
- Glimepiride as an active comparator to Sitagliptin (Active Comparator)
  Interventions: Drug: Sitagliptin; Drug: Glimepiride; Drug: Metformin; Drug: Insulin

INTERVENTIONS:
Drug: Sitagliptin — 100 mg once daily for 6 months
Drug: Glimepiride — 1 mg/2 mg/3 mg once daily
Drug: Metformin — >=1000 mg twice daily
Drug: Insulin — TDD > 10 IU once/twice daily

SUMMARY:
The purpose of the study is to determine the efficacy and safety of sitaglipin in the treatment of Type 2 diabetes mellitus (T2DM) patients with inadequate glycemic control using metformin and insulin.

DETAILED DESCRIPTION:
DPP-4 inhibitors enhance function of endogenous incretin that helps with glucose homoeostasis. DPP-4 inhibitors have been proved to promote glycemic control without increasing risk of hypoglycemia and weight gain. In addition, they may improve beta-cell function and do not have any known associations with overt cardiovascular or hepatic safety risks.

Addition of sitagliptin to treatment of T2DM patients poorly controlled on insulin +/- metformin has been shown to reduce HbA1c while being generally well-tolerated.

It could be clinically useful to add sitaglipin to treatment regimen of T2DM patients on stable therapy with insulin & metformin. Apart from glycemic reduction, secondary effects like prevention of weight gain, reduction in insulin dose, improved cardiovascular risk profile, etc. may be expected from addition of sitagliptin to treatment.

ELIGIBILITY:
Inclusion Criteria:

* T2DM patients on metformin and biphasic or basal regimens of insulin
* HbA1c ≥7.3% to ≤8.5%
* Age: 25 to 60 yrs
* Insulin TDD > 10 IU

Exclusion Criteria:

* Use of acarbose, pioglitazone or short-acting insulin analogues at time of run-in phase
* History of type 1 diabetes mellitus
* Creatinine clearance ≤50 mL/min
* Chronic liver & kidney diseases, SGOT/PT≥2.5x upper limit of normal, uncontrolled thyroid disorders , cardiac failure, hemochromatosis, autoimmune disorders, corticosteroid intake.
* BMI >40 kg/m2

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 440 (Actual)
Dates: Start 2012-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Reduction in HbA1c from baseline | six months
  To confirm the efficacy of metformin+ insulin+ sitagliptin in controlling glycemia with respect to change from baseline in HbA1c after 24 weeks of administration. This will be accomplished by comparing the difference in change from baseline in HbA1c after 24 weeks of administration, compared with metformin+insulin+glimepiride to a non-inferiority limit of 0.3% , and if non-inferiority is proven, to a superiority limit of 0%.

SECONDARY OUTCOMES:
Change in total daily dose (TDD) of insulin | 6 months
  Change from baseline in insulin TDD (30-day geometric mean) at Month 6
Episodes of hypoglycemia | 6 months
  Hypoglycemia (Total, severe, nocturnal) (From Month 0 to Month 6), as assessed by questionnaire and supplemented by SMBG values, if available
Proportion of patients with HbA1c reduction | 6 months
  Proportion of patients, who completed treatment , with HbA1c value <6.5% & ≤7.3% at end of study (Month 6)
change in weight and BMI | 6 months
Change in both HbA1c and TDD | 6 months
  Proportion of patients achieving both HbA1c ≤6.5% AND reduction in TDD (total daily dose of insulin)
Change in insulin resistance and beta cell function | 6 months
  Change from baseline in c-peptide levels, homeostasis model assessments of β-cell function and insulin resistance (HOMA-β and HOMA-IR)
Change in lipid profile from baseline | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jothydev Kesavadev, MD, Principal Investigator — Jothydev's Diabetes and Research Center
Locations (1):
- Jothydev's Diabetes and Research Center, Thiruvananthapuram, Kerala, India